CLINICAL TRIAL: NCT07001748
Title: Protocol EA2234: A Randomized Phase II/III Trial of Intraperitoneal Paclitaxel Plus Systemic Treatment vs Systemic Treatment Alone in Gastric Carcinomatosis - STOPGAP II
Brief Title: Testing the Addition of Paclitaxel Administered Into the Abdominal Cavity Combined With Chemotherapy for Patients With Gastric Cancer Spread to the Abdominal Cavity
Acronym: STOPGAP II
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA2234; U10CA180820 (NIH); NCI-2025-01831 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA2234 (Other: ECOG-ACRIN Cancer Research Group); EA2234 (Other: CTEP)
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Peritoneal Carcinomatosis
Keywords: EA2234; Intraperitoneal Paclitaxel; STOPGAP II; STOPGAP I; Gastric Carcinomatosis
MeSH Terms: conditions — Peritoneal Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Specimen Handling; Laparoscopy; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Step 1, Arm A (standard systemic therapy) (Active Comparator): Patients on Arm A will start systemic therapy with physician's choice of any standard-of-care systemic regimen for gastric/GEJ adenocarcinoma. Patients on Arm A will start systemic therapy as early as the day after Step 1 randomization and must start within 30 calendar days (including holidays) after Step 1 randomization. After 12 weeks (+/- 2 weeks) of standard of care treatment, patients will undergo a restaging assessment as outlined in Section 5.2 (restaging will occur at this timepoint, regardless of if the patient completed all 4 cycles or not). Patients who are found to have stable disease or a response may continue assigned standard of care treatment and will undergo restaging every 12 weeks (+/- 2 weeks) as outlined in Section 5.2. Treatment will continue until progression (radiographic progression or clinical progression as defined in Section 6), intolerance (unacceptable toxicity), or cytoreduction.
  Interventions: Drug: Standard of Care Chemotherapy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Diagnostic Laparoscopy; Procedure: Magnetic Resonance Imaging
- Step 1, Arm B (Systemic Therapy + Intraperitoneal Paclitaxel) (Experimental): Patients on Arm B will start systemic therapy + intraperitoneal paclitaxel as early as the day after Step 1 randomization and must start within 30 calendar days (including holidays) after Step 1 randomization.
  Therapy will be administered on Days 1 and 8 of a 21-day cycle for 4 cycles. After 12 weeks (+/- 2 weeks) of study treatment, patients will undergo restaging assessments as outlined in Section 5.2 (restaging will occur at this timepoint, regardless of if the patient completed all 4 cycles or not). Patients who are found to have stable disease or a response may continue assigned protocol treatment and will undergo restaging every 12 weeks (+/- 2 weeks) as outlined in Section 5.2. Treatment will continue until progression (radiographic progression or clinical progression as defined in Section 6), intolerance (unacceptable toxicity), or cytoreduction.
  Interventions: Drug: Standard of Care Chemotherapy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Diagnostic Laparoscopy; Procedure: Intraperitoneal Port Placement; Procedure: Magnetic Resonance Imaging; Drug: Intraperitoneal Paclitaxel

INTERVENTIONS:
Drug: Standard of Care Chemotherapy — The most common regimens are FOLFOX, CAPOX, FLOT, CF, and CX. Other local institutional standard of care regimens as well as targeted agents for gastric/GEJ adenocarcinoma are allowed.
  Other Names: best practice; standard of care; standard therapy
Procedure: Biospecimen Collection — Plasma is to be submitted at baseline and every three months for the first year or until progression, whichever comes first. For patients who have progression, their last plasma sample should be at time of progression.
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Restaging imaging with CT and/or diffusion weighted MRI with contrast will be obtained after completion of 12 weeks (+/- 2 weeks) of assigned treatment (restaging will occur at this timepoint, regardless of if the patient completed all 4 cycles or not). At this point, patients with stable disease or a response will continue assigned treatment. In the absence of radiological or clinical progression, if clinically indicated by treatment team, patients may undergo diagnostic laparoscopy to assess surgical candidacy at which time a PCI assessment and biopsies of peritoneal nodules, peritoneal lavage could be performed. Cytoreduction can be offered to patients with a PCI < 7 and if complete cytoreduction is feasible based on treating surgeon's discretion. If deemed a candidate for surgical cytoreduction, surgery should be performed within 6 weeks of the last study treatment in both arms.
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Diagnostic Laparoscopy — After induction of general anesthesia, administration of preoperative antibiotics and placement of appropriate laparoscopic ports, peritoneal lavage will be performed by instillation of 200 ml of normal saline in the left upper quadrant and allowed to dwell for 5 minutes after which it will be aspirated for cytology. Extent of peritoneal disease burden will be ascertained as per the Peritoneal Cancer Index (PCI) scoring system as outlined in Appendix V.
Procedure: Intraperitoneal Port Placement — Patients assigned to Arm B will undergo placement of indwelling tunneled intraperitoneal port with Teflon cuff following Step 1 randomization and during the diagnostic laparoscopy procedure.
  Arms: Step 1, Arm B (Systemic Therapy + Intraperitoneal Paclitaxel)
Procedure: Magnetic Resonance Imaging — Restaging imaging with CT and/or diffusion weighted MRI with contrast will be obtained after completion of 12 weeks (+/- 2 weeks) of assigned treatment (restaging will occur at this timepoint, regardless of if the patient completed all 4 cycles or not). At this point, patients with stable disease or a response will continue assigned treatment. In the absence of radiological or clinical progression, if clinically indicated by treatment team, patients may undergo diagnostic laparoscopy to assess surgical candidacy at which time a PCI assessment and biopsies of peritoneal nodules, peritoneal lavage could be performed. Cytoreduction can be offered to patients with a PCI < 7 and if complete cytoreduction is feasible based on treating surgeon's discretion. If deemed a candidate for surgical cytoreduction, surgery should be performed within 6 weeks of the last study treatment in both arms.
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Intraperitoneal Paclitaxel — Patients on Arm B will start systemic therapy + intraperitoneal paclitaxel as early as the day after Step 1 randomization and must start within 30 calendar days (including holidays) after Step 1 randomization as per the schedule shown in the table below.
  Therapy will be administered on Days 1 and 8 of a 21-day cycle for 4 cycles.
  Arms: Step 1, Arm B (Systemic Therapy + Intraperitoneal Paclitaxel)

SUMMARY:
This study is being done to answer the following questions:

Can we lower the chance of your gastric cancer from growing or spreading by administering paclitaxel chemotherapy directly into your abdominal cavity in addition to chemotherapy given through a vein in your arm? Will administering paclitaxel chemotherapy directly into your abdominal cavity, in addition to chemotherapy given through a vein in your arm help you live longer? We are doing this study because we want to find out if this approach is better or worse than the usual approach for your gastric cancer. The usual approach is defined as care most people get for gastric cancer.

If you decide to take part in this study, you will first receive a surgical procedure called a diagnostic laparoscopy. This will help the study doctors learn more about your gastric cancer. Laparoscopy is a minimally invasive surgery for which you will be placed under general anesthesia. Then the surgeon will make small incisions (5mm) on your belly through which a camera and thin instruments are introduced to evaluate the abdomen. This procedure takes about 1 hour to complete. Your study group will be assigned during the surgery. The study groups are described further in the 'What are the study groups?' section below.

If you are placed into the study group 1, you will not have an intraperitoneal port (a small device which is placed under the skin and fat of your upper abdomen and a tube that is placed into the abdomen).

If you are placed into the study group 2, you will have an intraperitoneal port placed. The reason is that in addition to standard chemotherapy, which is given through a vein in your arm, this port will be used to deliver the medication paclitaxel directly inside your abdomen when you are ready to start study treatment.

It is important to know that you will not know your study group until after the surgery is over. This is because information that is learned during the surgery will help determine which study group you are put in.

Once you have fully healed from this surgery, you will start study treatment. Depending on which study group you are assigned, you will either receive a standard chemotherapy regimen (the regimen will be chosen by you and your doctor) if you are in study group 1, or paclitaxel through a tube in your belly plus chemotherapy given through a vein in your arm if you are in study group 2. All participants will get treatment for three (3) months after which you will undergo reevaluation. If the disease is under control or responding to treatment, you may continue the assigned treatment until your disease gets worse, the side effects become too severe, or you may be offered a surgical procedure to remove the cancer if the amount of disease is low and can be completely removed as determined by a surgeon.

There is a very small chance that during the laparoscopy surgical procedure, the doctor might find something called "intra-abdominal adhesions". These are areas where the stomach has healed previously and created scar tissue. If this scar tissue prevents the surgeon from being able to place a port in the correct area, you would be ineligible to receive the study treatment. If this happens, you may still receive standard of care therapy after your surgery, but you will not be able to continue on the study. If you have more questions about this, you can ask your surgeon or the study team to help.

After you finish your study treatment, your doctor or study team will watch you for side effects. They will continue to follow your condition every three (3) months during the first two (2) years, then every six (6) months until year 5. You may be reevaluated with Chest/Abdomen/Pelvis scans every three-six (3-6) months for up to five (5) years if decided by your doctor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. In the phase II portion, to determine the progression free survival (PFS) from randomization.

II. In the phase III portion, to determine overall survival (OS) from randomization.

SECONDARY OBJECTIVE:

I. To compare the safety and tolerability of the intraperitoneal chemotherapy + systemic therapy regimen vs the systemic therapy alone regimen.

OUTLINE:

STEP 0: Patients undergo diagnostic laparoscopy within 4 weeks of study registration.

STEP 1: Patients are randomized to 1 of 2 arms at the time of Step 0 diagnostic laparoscopy.

ARM A: Patients receive standard of care systemic therapy per physician's choice. Patients with stable disease or a response after 12 weeks may continue to receive standard of care treatment in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection and computed tomography (CT) and/or magnetic resonance imaging (MRI) throughout the study and may undergo additional diagnostic laparoscopies as clinically indicated.

ARM B: Patients undergo placement of an intraperitoneal port. Patients receive leucovorin calcium intravenously (IV) over 15-30 minutes, fluorouracil IV push, paclitaxel IV over 1-2 hours and paclitaxel intraperitoneally (IP) on days 1 and 8 of each cycle. Cycles repeat every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients with stable disease or a response after 12 weeks may continue to receive treatment in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection and CT and/or MRI throughout the study and may undergo additional diagnostic laparoscopies as clinically indicated.

After completion of study treatment, patients are followed up every 3 months for 2 years then every 6 months for up to 5 years after Step 1 randomization.

ELIGIBILITY:
STEP 0 REGISTRATION:

* Patient must be at least 18 years of age
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Patient must have histologically or cytologically confirmed microsatellite stable (MSS) or mismatch repair (MMR) protein expression proficient primary gastric or gastroesophageal adenocarcinoma (Siewert 3) with synchronous cytology positive disease (cyt+) OR peritoneal carcinomatosis detected by imaging, laparoscopy or laparotomy. Patients with microsatellite instability-high (MSI-H/dMMR) mismatch repair deficient disease are not eligible
* Patient must have received a minimum of 3 months and a maximum of 6 months of first line systemic treatment
* Patient must be registered to Step 0 within 4 weeks of the last dose of first line systemic therapy. Patient must not have any ongoing significant adverse events that would prohibit them from undergoing a diagnostic laparoscopy procedure followed by further systemic and intraperitoneal therapy
* Patient must have no evidence of small or large bowel obstruction other than gastric outlet obstruction due to primary malignancy
* Patient must have no evidence of solid organ metastases except for ovarian metastases. Baseline imaging must be done within 30 days prior to Step 0 registration
* Patient must have no evidence of clinically significant radiologic peritoneal disease progression during first line systemic therapy
* Patient must have no evidence of extensive retroperitoneal lymph node metastases not amenable to resection during gastrectomy
* Patient must have no history of prior surgery that would preclude safe diagnostic laparoscopy and port placement
* Patient must have no evidence of massive ascites on imaging or history of two therapeutic paracentesis with drainage of more than 1.0 liter of ascites each time in 30 days prior to Step 0 registration
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better
* Patient must not have any uncontrolled intercurrent illness or any other significant condition(s) that would make this protocol unreasonably hazardous
* Patient must not have any known contraindications or drug allergies to the protocol treatment agents: paclitaxel, 5-fluorouracil, or leucovorin
* Leukocytes ≥ 2,000/uL (≤ 30 days prior to Step 0 registration)
* Absolute neutrophil count (ANC) ≥ 1,500/uL (≤ 30 days prior to Step 0 registration)
* Platelets ≥ 75,000/uL (≤ 30 days prior to Step 0 registration)
* Total bilirubin ≤ 1.5 institutional upper limit of normal (ULN). If patient has Gilbert's syndrome, total bilirubin must be < 2.0 mg/dL (≤ 30 days prior to Step 0 registration)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) ≤ 3.0 x institutional ULN (≤ 30 days prior to Step 0 registration)
* Creatinine clearance ≥ 30 mL/min (estimated using Cockcroft and Gault formula or measured) (≤ 30 days prior to Step 0 registration)
* Hemoglobin ≥ 8 g/dL (≤ 30 days prior to Step 0 registration)
* Serum albumin ≥ 2.5 g/dL (≤ 30 days prior to Step 0 registration)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of Step 0 registration are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used

  * All patients of childbearing potential must have a blood test or urine study within 14 days prior to Step 0 registration to rule out pregnancy
  * A patient of childbearing potential is defined as anyone, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Patient must not expect to conceive or father children by using accepted and effective method(s) of contraception (or by abstaining from sexual intercourse) for the duration of their participation in the study. Arm A patients must adhere to the contraceptive requirements outlined in the product specific package inserts while on protocol treatment. Arm B patients must continue contraceptive measures for at least 3 months after the last dose of protocol treatment. In addition, both Arm A and Arm B patients who continue with targeted agents must adhere to the contraceptive requirements outlined in the product specific package inserts while on protocol treatment
* Patient must have the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible

STEP 1 RANDOMIZATION:

* Patient must have undergone a diagnostic laparoscopy with peritoneal lavage performed and aspiration for cytology obtained
* The extent of peritoneal disease burden must have been assessed during the diagnostic laparoscopy with the Peritoneal Cancer Index (PCI) available
* Patient must not have extensive intraabdominal adhesions that preclude safe placement of the intraperitoneal port

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2030-05-30 (Estimated); Study Completion 2030-05-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (Phase II) | From randomization to progression or death without documentation of progression, assessed up to 5 years.
  For the Phase II portion, full information is expected to occur 12 months after accrual or 38 months after study activation. This power calculation is based on a stratified log rank test and accounts for a planned interim analysis at 50% information time. At 50% information time, futility test using Wieand rule would be conducted. If the study results show promising results for the investigational arm and reject the null hypothesis at interim efficacy analysis, the study will proceed to investigate Phase III portion without having a pause in accrual before starting Phase III. Otherwise, if the study is not futile at 50% information time (HR>1), then the study will proceed and wait for the data to reach 100% information, meaning that the study will wait until the data is mature for Phase II analysis (projected to wait 12 months after end of the accrual to collect 58 PFS events).
Overall survival (Phase III) | From randomization to the date of death, of any cause, assessed up to 5 years
  For the Phase III portion, a futility interim analysis is planned at 50% information time, projected to occur 4.3 years after study activation. However, because of the potential one year pause before starting Phase III portion, the futility interim analysis may occur early. Similar to the Phase II portion, the interim analysis for futility would use the Wieand rule to make sure the investigational arm is not doing worse than the control arm. For efficacy, interim analysis would start at 30% information time and be conducted every 6 months subsequently accordingly with the DSMC monitoring schedule. Approximately 1.5 additional years after completion of accrual, the OS analysis will reach 100% information time with 105 OS events.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 30 days after the last day of protocol treatment
  Safety and tolerability will be assessed by counting treatment-related grade 3 or higher toxicity events of the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Maheswari Senthil, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (10):
- United States (10):
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Irvine, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Orange, California
  - Schulze Family Foundation Cancer Clinic - Bonita Health Center, Bonita Springs, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Regional Cancer Center-Lee Memorial Health System, Fort Myers, Florida
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided